CLINICAL TRIAL: NCT02811757
Title: Clinical Outcomes After Arthroscopic Tenotomy or Tenodesis of the Long Head of the Biceps
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: CHU de Reims (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: PA13049
Record Dates: First submitted 2016-06-21; First posted 2016-06-23 (Estimated); Last update posted 2016-06-24 (Estimated); Status verified 2016-06

CONDITIONS: Arthroscopic Rotator Cuff
MeSH Terms: interventions — Tenotomy; Tenodesis

ARMS (2):
- tenodesis (Experimental)
  Interventions: Procedure: tenodesis
- tenotomy (Active Comparator)
  Interventions: Procedure: tenotomy

INTERVENTIONS:
Procedure: tenotomy
  Arms: tenotomy
Procedure: tenodesis
  Arms: tenodesis

SUMMARY:
Degenerative changes of the long head of the biceps brachii (LHB) are frequent and often associated with cuff tendinopathy. The function of the LHB in the shoulder is still controversial and uncertain, whereas its function in the elbow is certain. The biceps brachii is a flexor of the elbow and supinator of the forearm. Suppression of the pathologic long head of the biceps permits pain relief and is very reliable in the literature. Two options are available for the remaining tendon : simple tenotomy or tenodesis which consists to reattach the tendon to the humerus. Our hypothesis is that there is no difference in strength or endurance of the biceps brachii after tenotomy or tenodesis of the LHB. The aim of this study was to compare the strength and the endurance of the biceps brachii during supination and flexion after tenotomy or tenodesis of the LHB.

the investigators proposed a prospective and randomized study. All the patients treated in our department for an arthroscopic rotator cuff repair were included in this study after signed consent. Participants will complete isokinetic strength and endurance testing for elbow flexion and supination on the operative and nonoperative sides a minimum of 1 year after biceps tenotomy or tenodesis. The clinical evaluation included the range of motion measurement, Constant Score, Quick-DASH and SSV at 6 weeks, 3 months, 6 months and one year.

ELIGIBILITY:
Inclusion Criteria:

* surgery tenotomy or tenodesis type of the long head of the biceps (broken tendinopathy or not rotator cuff escaping a well conducted medical treatment and under a repair or cap pathology of the long head of the biceps during the arthroscopy)
* Patients treated in the orthopedic service of the Reims University Hospital
* Patients agreeing to participate in the research and who signed the informed consent
* Major patients.

Exclusion Criteria:

* prior Shoulder Surgery
* surgery scheduled contralateral shoulder
* patient protected by law

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2013-12; Primary Completion 2019-12 (Estimated)

PRIMARY OUTCOMES:
Max Peak Torque supination | 1 year
Max peak Torque Flexion | 1 year

CONTACTS AND LOCATIONS:
Locations (1):
- Chu Reims, France, Reims, France